CLINICAL TRIAL: NCT03370705
Title: A Multicentric Open-label Randomized Controlled Study for Evaluating the Improvement of Endothelial Function in Stage II Peripheral Arterial Obstructive Disease Patients Treated With Sulodexide + Conventional Treatment {CT] Vs CT Alone
Brief Title: Endothelial Function Evaluation in Patients With PAOD Treated With Sulodexide + Conventional Treatment (CT) Vs CT Alone
Acronym: AWAOMI2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alfa Wassermann Tunisia (Industry)
Collaborators: Poseidon CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP 12016 AW TN
Record Dates: First submitted 2017-11-24; First posted 2017-12-12 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Obstructive Disease
MeSH Terms: interventions — glucuronyl glucosamine glycan sulfate; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Atorvastatin; Platelet Aggregation Inhibitors; acetylsalicylic acid lysinate; Angiotensin-Converting Enzyme Inhibitors; Captopril

STUDY DESIGN:
Intervention Model Description: Randomized Multicentric open-label controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT group (Active Comparator): 78 patients will be treated by conventional treatment : antiplatelet therapy + ACE inhibitor +/- Statin in patients with cholesterol total level > 1,35 g/l
  Interventions: Drug: Statin; Drug: Antiplatelet Agents; Drug: ACE inhibitor
- Sulodexide + CT group (Experimental): 78 patients will be treated by :
  * Sulodexide (250ULS, twice daily , oral administration)
  * Conventional treatment : antiplatelet agents + ACE inhibitor +/- Statin in patients with cholesterol total level > 1,35 g/l
  Interventions: Drug: Sulodexide; Drug: Statin; Drug: Antiplatelet Agents; Drug: ACE inhibitor

INTERVENTIONS:
Drug: Sulodexide — Sulodexide 250 ULS twice daily per oral route
  Other Names: Vessel
  Arms: Sulodexide + CT group
Drug: Statin — Statin 20mg once daily per oral route,
  Other Names: Atorvastatin or equivalent
Drug: Antiplatelet Agents — Antiplatelet therapy 75mg once daily per oral route
  Other Names: lysine acetylsalicylate or equivalent
Drug: ACE inhibitor — ACE inhibitor 20mg once daily per oral route
  Other Names: Captopril or equivalent

SUMMARY:
A randomized Multicentric open-label controlled trial. The primary objective of the study is to assess the improvement of endothelial function under sulodexide + conventional treatment or conventional treatment alone in patients with Leriche-Fontaine stage II peripheral arterial obstructive disease (systolic ankle brachial index ABI < 0. 9).

DETAILED DESCRIPTION:
A randomized Multicentric open-label controlled trial. The primary objective of the study is to assess the improvement of endothelial function under sulodexide + conventional treatment (antiplatelet therapy; plus ACE inhibitor; plus Statin in patients with cholesterol total level > 1,35 g/l) or conventional treatment alone in patients with Leriche-Fontaine stage II peripheral arterial obstructive disease (systolic ankle brachial index ABI < 0. 9).

Criteria for efficacy evaluation are the assessement of the improvement of the Digital Thermal monitoring between base line (day 1) and day 180 measured by Vendys® and the measurement of the correlation between the Digital Thermal monitoring and the following parameters at base line, day 90 and day 180:

* Von Willebrand factor blood level.
* Clinical assessment as per pain free walking distance and maximum walking distance, as measured by walking machine.
* Fibrinogen blood level. Also an assessment of the study medication observance (patient's compliance) will be done.

Safety assessment will be done through the collection of the adverse events occurred during the study.

ELIGIBILITY:
Inclusion Criteria:

* Intermittent claudication.
* A systolic ankle brachial index ABI < 0. 9
* An age of over 40 years
* At least one cardiovascular risk factor (active or weaned Smoking, diabetes mellitus, hypertension, lipid disorders, obesity, and erectile dysfunction) or a history of coronary artery disease or transient ischemic stroke or established.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

* withdrawal of informed consent
* participation in another clinical trial with investigational drugs within the last 12 weeks or during the present trial period
* history of hypersensitivity to the investigational/conventional drugs
* Non claudicating patients and patients with critical ischemia
* Arteritis of non-atherosclerotic origin
* Patients treated with the oxalate or Naftidrofuryl Pentoxifiline Cilostazol or within 3 months that preceded the inclusion
* Patients receiving other agents that alter the secretion of NO (such as Sildenafil and Tadalafil) less than 2 weeks before inclusion
* Patients receiving a regimen based on nitrates or molsidomine or Bosentan
* Patients receiving Anti Vitamin K medication (AVK)
* Hemorrhagic accident dating less than 15 days before inclusion
* Heparin treatment or any treatment by low molecular weight heparins during the study for a continuous period of more than 10 days or a cumulative time during the study for more than 21 days.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2019-01-31 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline endothelial function after 6 months | between base line (day 1) and day 180
  Assess the improvement of the Digital Thermal monitoring measured by Vendys®: evaluation of the improvement of Fingertip Digital Thermal Monitoring (DTM) and the detection of a significant change of the FT2 parameters as per Endothelix discriminative values provided by the manufacturer between day 1 and day 180 (±15 days).

SECONDARY OUTCOMES:
Metric change of the walking distance | base line, day 90 and day 180:
  Metric variation of the walking distance: Clinical assessment as per pain free walking distance and maximum walking distance, measured by walking machine. A significant change for more than 30% of the walking distance at the assessment point, to consider it an improvement while analysing.
Change in Von Willebrand Factor (VWF) level | base line, day 90 and day 180
  Evidence of significant change in VWF level: Serum levels of Von Willebrand Factor will be measured by immunoturbidiometric method. An improvement of the level of VWF blood level by at least 10% in 1st assessment and 30% in last assessment compared to baseline values
Assessment of the study medication observance patient's compliance | 180 days
  Compliance will be stated in accordance to the results stated by the patients during remote monitoring at days, 30, 80, 170, and the drug accountability performed by doctors at days 90 and 180. It will be measured in % of the total destined dose expressed in number of intakes and days of treatment.
Assessment of safety | 180 days
  Safety will be assessed by checklist questioning during visits and remote interactions, investigators will be responsible for collection and notification to the Sponsor and authorities in case of Serious Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Imed Frikha, MD, Principal Investigator — STCCV
Locations (3):
- Tunisia (3):
  - InvSite Poseidon0031, Sfax
  - InvSite Poseidon 0022, Sousse
  - InvSite Poseidon0011, Tunis

IPD SHARING:
Plan to Share IPD: Undecided